CLINICAL TRIAL: NCT04104165
Title: Intermittent Versus Continous Catheterization for Treatment of Postpartum Urinary Retention.
Brief Title: Treatment of Postpartum Urinary Retention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Principal Investigator, ROY LAUTERBACH MD, Principal investigator, Rambam Health Care Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0515-19-RMB
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2022-08-16 (Actual); Status verified 2022-08

CONDITIONS: Retention, Urinary
MeSH Terms: conditions — Urinary Retention

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intermittent catheterization (Active Comparator): women who are catheterized intermittently every 6-8 hours up to a total time of 48 hours
  Interventions: Device: Foley Catheter
- Continous catheterization (Active Comparator): women which will have an indwelling catheter inserted for 24 hours
  Interventions: Device: Foley Catheter

INTERVENTIONS:
Device: Foley Catheter — Foley catheter used for treatment of urinary retention

SUMMARY:
The aim of the study is to evaluate what is the most effective catheterization duration to resolve covert and overt postpartum urinary retention following vaginal delivery and caesarean delivery, with the highest patients' satisfaction.

DETAILED DESCRIPTION:
1. Women who are unable to micturate for more than 6-8 hours following vaginal delivery or within six to eight hours following removal of an indwelling catheter after cesarean delivery (overt postpartum urinary retention), or women with postvoid residual bladder volume of at least 150 mL (covert postpartum urinary retention) will be randomized into 2 groups: one group will include women who are catheterized intermittently every 6-8 hours up to a total time of 48 hours. If at any time, post voiding residual volume is less than 150cc (assessed by ultrasound or by catheterization), no additional catheterization is needed. The second group will include women which will have an indwelling catheter inserted for 24 hours. The catheter will be removed 24 hours following its insertion and post voiding residual volume will be assessed 6 hours following the catheter removal (by ultrasound or by catheterization). In cases of post voiding residual volume more than 150 cc or women are unable to micturate spontaneously, an indwelling catheter will be inserted for additional 24 hours.
2. After 48 hours from postpartum urinary retention diagnosis, an indwelling catheter will be inserted for additional time that will be set at every center by its common protocol.

ELIGIBILITY:
Inclusion Criteria:

* Women who deliver at one of the centers included in the study
* Overt postpartum urinary retention which refers to the absence of spontaneous micturition within six to eight hours of vaginal delivery; or within six to eight hours following removal of an indwelling catheter after cesarean delivery
* Covert postpartum urinary retention diagnosed by ultrasound or catheterization of more than 150cc

Exclusion Criteria:

* Spontaneous micturition 6-8 hours following vaginal or cesarean delivery
* postpartum urinary retention less than 150cc on ultrasound
* Known urinary tract infection

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female patients
Enrollment: 146 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Mean time for urinary retention resolution. | Up to 10 days from diagnosis
  Mean time for urinary retention resolution following the intervention.

SECONDARY OUTCOMES:
Urinary tract infection rate | Up to 96 hours from diagnosis
  Incidence of Urinary tract infections
Length of hospital stay | Up to 96 hours from diagnosis
  Length of hospital stay

CONTACTS AND LOCATIONS:
Overall Officials: Roy Lauterbach, MD, Principal Investigator — Rambam Healthcare Campus
Locations (1):
- Rambam Healthcare Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No